CLINICAL TRIAL: NCT00928746
Title: ATROVENT HFA Actuation Indicator Open-Label Study in Adults With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Actuation Indicator Trial in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Purpose: Treatment
Other Study IDs: 244.2507
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2010-09-28 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (1):
- ATROVENT 42mcg (Other)
  Interventions: Device: Ipratropium bromide

INTERVENTIONS:
Device: Ipratropium bromide

SUMMARY:
The primary objective of this study is to evaluate the performance, accuracy, and handling of the actuation indicator in patients with COPD. The actuation indicator is integrated into mouthpiece of the ipratropium bromide HFA inhalation aerosol device. As part of Boehringer Ingelheim's program to qualify an actuation indicator for use with the ipratropium bromide HFA inhalation aerosol device, this study is intended to complement the results from the ongoing in-vitro studies.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of COPD based on medical history at a severity to require maintenance treatment with a bronchodilator
2. Male or female patients 40 years of age or older
3. A smoking history of more than ten pack-years. A pack-year is defined as the equivalent of smoking one pack of 20 cigarettes per day for a year
4. Must be able to use the study MDI with the mouthpiece containing actuation indicator

Exclusion Criteria:

1. Significant diseases other than COPD are excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
2. Malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last three months. Patients with treated basal cell carcinoma are allowed
3. History of asthma
4. Significant history active alcohol or drug abuse
5. Known active tuberculosis
6. Known narrow-angle glaucoma
7. Current significant psychiatric disorders
8. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e., oral contraceptives, intrauterine devices or diaphragm with spermicide, or Norplant®)
9. Known hypersensitivity to anticholinergic drugs, any other component of the ipratropium bromide, HFA-134a or MDI components
10. Previous participation in this trial
11. Patients who are currently participating in another trial and/or who have received investigational drug within the past 30 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (7):
- United States (7):
  - 244.2507.0107 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 244.2507.0106 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 244.2507.0102 Boehringer Ingelheim Investigational Site, Gaffney, South Carolina
  - 244.2507.0104 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 244.2507.0105 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 244.2507.0103 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 244.2507.0101 Boehringer Ingelheim Investigational Site, Union, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- ATROVENT 42mcg: ATROVENT HFA (42 mcg)- Oral inhalation
Period: Overall Study
Arm/Group | ATROVENT 42mcg
Started | 142
Completed | 136
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Patients who were entered into this study and documented to have taken at least one dose of study medication (treated set).
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 77
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 20
  White | 122
Alcohol status [Number; unit: participants]
  Does not drink alcohol | 94
  Drinks alcohol - should not interfere with trial | 48
Smoking history [Number; unit: participants]
  Ex-smoker | 62
  Currently smoke | 80
Height [Mean (Standard Deviation); unit: centimeters] | 167.2 (15.7)
Weight [Mean (Standard Deviation); unit: kilograms] | 88.8 (27.7)

OUTCOME MEASURES:

1. Primary Outcome: Actuations Registered by the Actuation Indicator
Description: This outcome measure presents the number of actuations (doses) of medication used in the specific time frame as measured by the actuation indicator
Time Frame: 21 Days
Population: The primary analysis was performed using the Full Analysis Set (FAS).
Measure: Median (Standard Deviation); unit: Count
Groups:
- ATROVENT 42mcg: ATROVENT HFA (42 mcg- Oral inhalation) - 180 Actuations group
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
Count | 167 (19.44)

2. Primary Outcome: Actuations Dispensed
Description: Actuations dispensed is determined by the weight differential of the canister over the course of the study divided by the shot weight
Time Frame: 21 Days
Population: The primary analysis was performed using the Full Analysis Set (FAS)
Measure: Median (Standard Deviation); unit: Count
Groups:
- ATROVENT 42mcg: ATROVENT HFA (42 mcg - Oral inhalation) - 180 Actuations group
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
Count | 159.77 (20.78)

3. Primary Outcome: Difference Between the Number of Actuations Registered by Actuation Indicator Versus Actuations Dispensed
Description: Difference between the number of actuations registered by the actuation indicator and the number of actuations dispensed (calculated using weight differential and shot weight)
Time Frame: 21 Days
Population: The primary analysis was performed using the Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Count
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
Count | 1.85 (9.8) [1.29 to 2.90]

4. Secondary Outcome: Actuations Recorded on Patient Diary
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Median (Standard Deviation); unit: Count
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
Count | 168 (20.57)

5. Secondary Outcome: Actuations Based on Advancing the Actuation Indicator
Description: Actuations based on advancing the actuation indicator to a zero reading or to the next increment
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Median (Standard Deviation); unit: Count
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 121
Count | 166 (19.57)

6. Secondary Outcome: Actuations Registered by the Actuation Indicator and Read by Site Coordinator
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Median (Standard Deviation); unit: Count
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
Count | 164 (19.66)

7. Secondary Outcome: Difference Between the Number of Actuations Recorded on Patient Diary Versus Actuations Dispensed
Description: Difference between the number of actuations recorded on patient diary and the number of actuations dispensed (calculated using weight differential and shot weight)
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: Count
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
Count | 5.07 (18.85) [3.11 to 8.54]

8. Secondary Outcome: Difference Between the Number of Actuations Based on Advancing Actuation Indicator Versus Actuations Dispensed
Description: Difference between the number of actuations based on advancing the actuation indicator to a zero reading or to the next increment and the number of actuations dispensed (calculated using weight differential and shot weight)
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: Count
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 121
Count | 1.71 (9.3) [0.18 to 3.84]

9. Secondary Outcome: Difference Between the Number of Actuations Registered by the Actuation Indicator and Read by Site Coordinator Versus Actuations Dispensed
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: Count
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
Count | 3.33 (9.8) [2.06 to 4.35]

10. Secondary Outcome: Number of Participants Who Reported Problems With Use of Inhaler With Integrated Dose Counter According to Patient Handling Questionnaire
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Number; unit: participants
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
participants
  No | 113
  Yes | 11

11. Secondary Outcome: Number of Participants Who Reported Problems With Seeing Red Warning Indicating Inhaler Near End of Recommended Doses According to Patient Handling Questionnaire
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Number; unit: participants
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
participants
  no | 15
  yes | 109

12. Secondary Outcome: Number of Participants Who Reported Problems With Inhaler and Dose Counter Performing as Expected Based on Instructions According to Patient Handling Questionnaire
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Number; unit: participants
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
participants
  No | 5
  Yes | 119

13. Secondary Outcome: Number of Participants Who Reported Satisfaction With Performance of the Dose Counter for Indicating Approximately How Many Doses Remain in Inhaler According to Patient Handling Questionnaire
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Number; unit: participants
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
participants
  No | 6
  Yes | 118

14. Secondary Outcome: Number of Participants Who Reported Satisfaction That the Dose Counter Worked Reliably According to Patient Handling Questionnaire
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Number; unit: participants
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
participants
  No | 6
  Yes | 118

15. Secondary Outcome: Number of Participants Who Reported Satisfaction With Ease of Use of the Dose Counter According to Patient Handling Questionnaire
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Number; unit: participants
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
participants
  No | 3
  Yes | 121

16. Secondary Outcome: Number of Participants Who Reported Satisfaction With Dose Counter in the Mouthpiece of the Inhaler According to Patient Handling Questionnaire
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Number; unit: participants
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
participants
  No | 4
  Yes | 120

17. Secondary Outcome: Number of Participants Having Any Additional Comments According to Patient Handling Questionnaire
Time Frame: 21 Days
Population: This secondary analysis was performed using the Full Analysis Set (FAS).
Measure: Number; unit: participants
Arm/Group | ATROVENT 42mcg
Number analyzed (Participants) | 124
participants
  No | 103
  Yes | 21

ADVERSE EVENTS:
Time Frame: Up to 21 days
Arm/Group | ATROVENT 42mcg
Serious Adverse Events (participants affected / at risk) | 2/142
Other Adverse Events (participants affected / at risk) | 0/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATROVENT 42mcg (N=142)
Loss of consciousness (Nervous system disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.